CLINICAL TRIAL: NCT01122732
Title: Comparison of Pain Relief After US Guided Non Stimulating Interscalene Catheter Placement vs Stimulating Catheter Placement in Total Shoulder Arthroplasty;a Randomized Study
Brief Title: Comparison of Pain Relief After Non Stimulating Interscalene Catheter Placement vs Stimulating Catheter Placement in Total Shoulder Arthroplasty.
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 10-242-B
Record Dates: First submitted 2010-05-11; First posted 2010-05-13 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Pain; Shoulder; Arthroplasty
Keywords: nerve block; continuous catheter; shoulder surgery; pain control after total shoulder arthroplasty
MeSH Terms: conditions — Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- US Group: Interscalene catheter will be placed with US guidance without any nerve stimulation guidance.
- NS Group: Catheter will be placed using nerve stimulation guidance

SUMMARY:
1. Interscalene continuous catheter is a very effective way of controlling pain in total shoulder arthroplasty. To ensure proper placement, nerve stimulating catheter is quite often used.
2. Ultrasound can help proper placement of catheter without relying on nerve stimulation.
3. The plan of the study is to compare two techniques head to head to see if they are equally effective or one is better than others.

DETAILED DESCRIPTION:
After consent patients will be randomized to one of the two groups: Control Group or the Experimental Group. Patients will be blinded to the group assignment. As both catheters are placed using almost the same technique, the subjects will be unable to tell type of catheter they will be getting..

Every procedure will be done after starting intravenous access and placing standard anesthesia monitors (EKG, Blood Pressure Cuff and Pulse-Ox) on the patients. For comfort care sedation will be titrated using accepted American Society of Anesthesiology and American society of Regional Anesthesia Guidelines.

In the Control Group the patient will have interscalene catheter placed using nerve stimulation technique. Initially ultrasound guidance will be used to visualize brachial plexus at the cricoid level with the intent to visualize upper trunks or roots. Then following established guidelines a nerve stimulating catheter will be placed. This will be done using an ARROW NERVE KIT. The kit is FAD approved for this purpose.. Following accepted aseptic guidelines the nerves will be visualized at the base of the neck using ultrasound machine. Once proper nerve roots or trunks visualized, kit provided 17gauge insulated Touhy needle will be used to access the brachial plexus. Once twitches elicited in Deltoid, biceps or triceps muscles at 0.5 mamp, catheter will be threaded via the needle while maintaining twitch at 0.5 mamp or less. Once catheter is threaded 3 cm beyond the tip, Touhy needle will be removed. Catheter will be tested for proper placement using lidocaine and epinephrine as is recommended by Regional Anesthesia Society guidelines. Thereafter 3 mg/kg of 0.5 % bupivacaine will be injected in small blouses via the catheter.

In the Experimental Group, after placement of monitors, the nerves will be visualized using ultrasound machine. Once nerve visualized at the cricoids level, proper tip of Touhy needle will be guided using hydro-dissection technique. Once in good place, catheter will be threaded 3 cm into the space. They subjects will be dosed using 0.5% bupivacaine 3 mg/kg for the surgery via the catheter. Adequacy of catheter placement will be judged by examining the spread of local anesthetics around the plexus.

The extent of block before the surgery will be evaluated at 30 minutes post injection. Surgery will be done with sedation. Conversion of anesthetic technique to general anesthesia will be considered failure of the technique to provide adequate surgical anesthesia.

At the end of the case the patient will be taken to recovery and will be evaluated for pain. If patient is having pain of 3 or more then they will be treated as follows.

In each catheter group patient will be dosed with 10 ml 1% lidocaine. If it fails to provide any relief then the catheter will be pulled back and another 10 ml1% lidocaine will be given. If still not effective then it will be replaced. Refusal of patient to replace the catheter will result in pt dropping out of the study.

Working catheter will be left in place for at least 48 hrs. Patients will be allowed to take oral pain medicines as prescribed by their surgeons. The patient will be sent home with pain pump to continuously give them 0.125% bupivacaine at 5 ml per hr with an option to get extra dose of 5 ml every one hr if needed. The pain control will be monitored while in-house and by phone daily till catheter comes out.

ELIGIBILITY:
Inclusion Criteria:

* 18 yr or older
* patient agreed to continuous regional block

Exclusion Criteria:

* minor
* patient refusal
* any neuropathy
* allergies to local anesthetic,
* inability to obtain informed consent for any reason, Opioid user, chronic pain patients or unanticipated procedure other than total shoulder arthroplasty

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all subjects having total shoulder arthroplasty.
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2010-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Pain | 2-3 days after surgery
  Pain will be monitored over the next 2-3 days while subjects have catheter inplace. Sleep, total oral analgesic intake will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: TARIQ MALIK, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago Hospitals, Chicago, Illinois, United States